CLINICAL TRIAL: NCT03952000
Title: Influence of Prior Walking on Endothelial Function and Coronary Heart Disease Risk Markers in Centrally Obese South Asian and White European Men
Brief Title: Influence of Prior Walking on Postprandial Metabolism in Centrally Obese Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Principal Investigator, Matthew Roberts, Principal investigator, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R18-P120
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases; Endothelial Dysfunction; Insulin Resistance; Oxidative Stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Exercise (Experimental): Exercise: Participants will walk for 60 minutes at 60% maximal oxygen uptake on day 1.
  Interventions: Behavioral: Exercise
- No Intervention: Control (No Intervention): Participants will rest on day 1.

INTERVENTIONS:
Behavioral: Exercise — A 60 minute walk at 60% maximal oxygen uptake.
  Arms: Experimental: Exercise

SUMMARY:
The present study will investigate the effect of prior walking on postprandial metabolism and endothelial function in centrally obese South Asian and White European men.

Participants will complete two, 2-day trials in a random, crossover design separated by at least a week.

On day 1, participants will either rest or complete a 60 minute walk at 60% maximal oxygen uptake. On day 2, participants will arrive at 08:00 having fasted overnight and a baseline venous blood sample and endothelial function measurement will be taken. Participants will consume a high-fat breakfast and lunch and 12 subsequent venous blood samples will be taken throughout the day at standardised intervals to measure a variety of coronary heart disease risk markers. A second endothelial function measurement will be completed 2 hours after the breakfast. Blood pressure will be measured every hour.

It is expected that the South Asian participants will have impaired metabolism and endothelial function compared to their European counterparts but the bout of exercise performed on day 1 will mitigate these responses.

DETAILED DESCRIPTION:
South Asians have a higher-than-average risk of coronary heart disease. The reasons for this are unclear, but physical inactivity and/or poor responsiveness to exercise may play a role. It is important to understand the effect of exercise on endothelial function and coronary heart disease risk markers in the hope that exercise can be prescribed as an effective treatment to mitigate endothelial dysfunction and the risk of heart disease.

Previous research from the investigators' laboratory has indicated that postprandial metabolism is impaired in South Asian men, but this, and other coronary heart disease risk markers, can be improved with acute exercise. However, the previous research was conducted in apparently healthy South Asian and White European men. The investigators now wish to quantify and compare the coronary heart disease risk marker and endothelial function response to acute exercise in centrally obese South Asian and White European individuals who are at a higher risk for diabetes and cardiovascular disease.

On visit 1, participants will attend the laboratory to undergo preliminary assessments and to be familiarised with the laboratory environment and study procedures. Specifically, health status, habitual physical activity, dietary habits and anthropometric data (height, weight, waist and hip circumference, body fat) will be collected. A HbA1c test will be performed to check participants are not diabetic. The modified Bruce Treadmill test will be performed to predict maximal oxygen uptake.

On visit 2, participants will undergo a magnetic resonance imaging (MRI) scan to quantify regional body composition comprising abdominal subcutaneous adipose tissue, visceral adipose tissue, liver fat percentage, thigh intramuscular adipose tissue and thigh muscle volume.

On visits 3-6 participants will complete two, 2-day trials in a random, crossover design separated by at least 1 week. On day 1 of both trials, participants will arrive fasted at 08:00 and a baseline blood sample, blood pressure and endothelial function measurement will be taken. Participants will consume a standardised high fat breakfast at 09:00 and lunch at 13:00. At 15:30 the participants will walk for 60 minutes at 60% maximal oxygen uptake and complete a second endothelial function measurement at 16:45. Participants will leave the laboratory with a standardised evening meal to consume before 22:00. The control trial will be the same, except no exercise will be performed.

On day 2, participants will arrive at 08:00 having fasted overnight for 10h (except plain water). A cannula will be inserted into the antecubital vein for collection of venous blood samples. Blood pressure will be measured at 08:00 (0h) and again at hourly intervals throughout the day. Endothelial function will measured at 08:15 (0.25h) and again at 3h. At 0h, a fasting blood sample will be collected. Subsequent venous blood samples will be collected at 1.5, 1.75, 2, 3, 4, 5, 5.5, 5.75, 6, 7, 8 and 9h. Participants will consume a standardised high fat breakfast at 1h and a standardised high fat lunch at 5h. The meals consist of 57% fat, 32% carbohydrate and 11% protein. The meals provide 14.3 kcal per kg of body mass.

Participants will rest in the laboratory throughout day 2 of both the exercise and control trials.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 year old South Asian and White European men;
* Centrally obese (waist circumference >90cm for South Asians, >94cm for White Europeans);
* Weight stable for the past 3 months;
* Non-smokers;
* No known contradictions to maximal exertion exercise.

Exclusion Criteria:

* Musculoskeletal injury that has affected normal ambulation within the last month;
* Congenital heart disease;
* Any muscle or bone injuries that do not allow them to walk on a treadmill;
* Uncontrolled exercise-induced asthma;
* Coagulation or bleeding disorders;
* Diabetes (metabolism will be different to non-diabetics potentially skewing the data);
* Taking any medication that might influence fat metabolism;
* Taking any medication that might influence blood glucose (e.g., insulin for diabetes);
* Heart conditions;
* Smoking;
* Dieting or restrained eating behaviours;
* Weight fluctuation greater than 3 kg in the previous 3 months to study enrolment;
* A food allergy.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Triacylglycerol changes in response to exercise and feeding | Day 1 fasting. Day 2 fasting (0 hour point), 1.5hours, 1.75hours, 2hours, 3hours, 4hours, 5hours, 5.5hours, 5.75hours, 6hours, 7hours, 8hours and 9hours.
  Fasting on day 1 and 2. Time-course of plasma triacylglycerol concentrations in response to exercise and/or feeding on day 2.
Endothelial function changes in response to exercise and feeding | Day 1 fasting and 8.75hours. Day 2 fasting and 2.5hours.
  Changes in endothelial function via flow-mediated dilatation in response to feeding and exercise.

SECONDARY OUTCOMES:
Glucose changes in response to exercise and/or feeding | Day 1 fasting. Day 2 fasting (0 hour point), 1.5hours, 1.75hours, 2hours, 3hours, 4hours, 5hours, 5.5hours, 5.75hours, 6hours, 7hours, 8hours and 9hours.
  Fasting on day 1 and 2. Time-course of plasma glucose concentrations in response to exercise and/or feeding on day 2.
Blood pressure changes in response to exercise and/or feeding | Day 1 fasting. Day 2 fasting (0 hour point) and 1hours, 2hours, 3hours, 4hours, 5hours, 6hours, 7hours, 8hours and 9hours.
  Changes in blood pressure (systolic and diastolic).
Total cholesterol | Day 1 fasting. Day 2 fasting.
  Fasting plasma total cholesterol on day 1 and day 2 of both trials.
Insulin changes in response to exercise and/or feeding | Day 1 fasting. Day 2 fasting (0 hour point), 1.5hours, 2hours, 4hours, 5hours, 5.5hours, 7hours, 8hours.
  Fasting on day 1 and 2. Time-course of plasma insulin concentrations in response to exercise and/or feeding on day 2.
High-density lipoprotein cholesterol | Day 1 fasting. Day 2 fasting.
  Fasting high-density lipoprotein cholesterol on day 1 and 2 of both trials.
Low-density lipoprotein cholesterol | Day 1 fasting. Day 2 fasting.
  Fasting low-density lipoprotein cholesterol on day 1 and 2 of both trials.
Non-esterified fatty acids changes in response to exercise and/or feeding | Day 1 fasting. Day 2 fasting (0 hour point), 1.5hours, 2hours, 4hours, 5hours, 5.5hours, 7hours and 9hours.
  Fasting on day 1 and 2. Time-course of plasma non-esterified fatty acid concentrations in response to exercise and/or feeding on day 2.
Interleukin-6 changes in response to exercise and/or feeding | Day 1 fasting. Day 2 fasting (0 hour point), 3hours, 6hours and 8hours.
  Fasting on day 1 and 2. Time-course of plasma interleukin-6 concentrations in response to exercise and/or feeding on day 2.
C-Reactive protein changes in response to exercise and/or feeding | Day 1 fasting. Day 2 fasting (0 hour point), 3hours, 6hours and 8hours.
  Fasting on day 1 and 2. Time-course of plasma C-Reactive protein concentrations in response to exercise and/or feeding on day 2.
Tumor Necrosis Factor concentrations | Day 1 fasting. Day 2 fasting.
  Fasting tumor necrosis factor on day 1 and 2 of both trials.
Peroxiredoxin-4 changes in response to exercise and/or feeding | Day 1 fasting. Day 2 fasting (0 hour point), 3hours, 6hours and 8hours.
  Fasting on day 1 and 2. Time-course of plasma peroxiredoxin-4 concentrations across day 2 of both trials.
Superoxide dismutase 3 | Day 1 fasting. Day 2 fasting (0 hour point), 3hours, 6hours and 8hours.
  Fasting on day 1 and 2. Time-course of plasma Superoxide dismutase 3 concentrations across day 2 of both trials

CONTACTS AND LOCATIONS:
Overall Officials: David Stensel, Principal Investigator — Loughborough University
Locations (1):
- National Centre for Sport and Exercise Medicine, Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data for all primary and secondary outcome measures will be made available upon request. Study protocol, statistical analysis plan and informed consent forms are also available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available in 6 months after publication for 1 year.
Access Criteria: Data will be available to other researchers who would like to run the same statistical methods we have used to check the interpretation of results.

REFERENCES:
- [Background] Arjunan SP, Deighton K, Bishop NC, King J, Reischak-Oliveira A, Rogan A, Sedgwick M, Thackray AE, Webb D, Stensel DJ. The effect of prior walking on coronary heart disease risk markers in South Asian and European men. Eur J Appl Physiol. 2015 Dec;115(12):2641-51. doi: 10.1007/s00421-015-3269-7. Epub 2015 Oct 5. PMID 26438068
- [Background] Arjunan SP, Bishop NC, Reischak-Oliveira A, Stensel DJ. Exercise and coronary heart disease risk markers in South Asian and European men. Med Sci Sports Exerc. 2013 Jul;45(7):1261-8. doi: 10.1249/MSS.0b013e3182853ecf. PMID 23470315